CLINICAL TRIAL: NCT05941780
Title: Pain Phenotypes in Patients with Fibromyalgia Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Director, Kutahya Health Sciences University
Other Study IDs: painclassificationFMS
Record Dates: First submitted 2023-06-22; First posted 2023-07-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia, Primary; Fibromyalgia; Chronic Pain Syndrome; Pain, Neuropathic; Nociceptive Pain; Central Sensitisation
MeSH Terms: conditions — Fibromyalgia; Neuralgia; Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Pain classification method — A current clinical algorithm will be used to determine the predominant type of pain in individuals with FMS. The classification to diagnose nociceptive, neuropathic and nociplastic pain will based on a recent method developed by Nijs et al. This method consists of seven steps in total. These steps question the following, respectively: duration of pain, pain distribution, presence of nociceptive pain, presence of neuropathic pain, phenomenon of hypersensitivity, presence of hypersensitization and presence of specific comorbidity. Besides, inter-rater and intra-rater reliability of pain classification algorithm will be determined by two independent researchers.

SUMMARY:
Fibromyalgia Syndrome (FMS); is a complex syndrome characterized by many symptoms such as chronic widespread pain, fatigue and sleep disorders, cognitive dysfunctions and psychiatric disorders. It has been stated that there is an urgent need for studies examining the clinicimetric and psychometric properties of the pain phenotype criteria in terms of patients receiving the most appropriate treatment, clinicians deciding on the appropriate treatment, and contributing to the research of scientists. Despite all this, no study has yet been found that describes the pain phenotypes in fibromyalgia syndrome and how different types of pain affect patients.

The primary aim of this study is to determine the chronic pain phenotypes in individuals with FMS. The secondary aim of this study to determine the inter-rater and intra-rater reliability of the algorithm used in the determination of pain phenotypes and to assessment the clinical effects of different pain phenotypes on individuals with FMS in terms of pain severity, disease severity, quality of life and catastrophe.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with fibromyalgia syndrome according to the criteria of the American Rheumatology Association ,
* not receiving active treatment related to physiotherapy,
* volunteering to participate in the study

Exclusion Criteria:

* diagnosed endocrine, neuromuscular, infectious and inflammatory diseases,
* severe mental and psychological disorders, using psychological drugs (SSRIs and SNRIs)
* illiterate
* problems with hearing and vision

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Participants meeting the inclusion criteria will be taken for this cross-sectional study. Individuals with FMS who apply to Pamukkale University Rheumatology Clinic will be screened for eligibility by their clinic physicians and will then be asked to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative sensory test: static tactile mechanical threshold | 10 minutes
  Von Frey Monofilaments (2 gr- 26 gr) will be used assessment for the static tactile mechanical detection threshold.
Quantitative sensory test: hot-cold pain threshold | 5 minutes
  Coins will be used for the hot-cold pain threshold. The cold sensing test will be done with a coin held at room temperature. The hot sensing test will be done in the form of a coin placed in the pocket and applied to the participant after waiting for 30 minutes.
Quantitative sensory test: static mechanical allodynia | 5 minutes
  A digital algometer device (JTech) will be used for static mechanical allodynia (pressure pain threshold). In the device, the pain sensation will be tested by applying 4 kg of pressure to the participant.
Quantitative sensory test: dynamic mechanical allodynia | 5 minutes
  A soft brush will be used for dynamic mechanical allodynia. The brush will be gently moved over the skin at a speed of 3-5 cm per second in a fixed direction over the patients primary painful area.
Quantitative sensory test: vibration sense | 5 minutes
  128 Hz tuning fork will be used in vibration assessment. The device will be applied over the bony prominences in the painful area of the patient.
Margolis Pain Diagram | one minute
  The Margolis Pain Diagram, consists of a dorsal and a ventral drawing body, is used to assess the location and distribution of the pain [20]. Participants will ask to point out the place where they experience pain during the preceding 4 weeks for at least 24 hours.
Numeric pain rating scale | one minute
  The NPRS was used to assess the participants' pain levels. In the NPRS, patients are asked to verbally rate the severity of their pain on a scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Revised Fibromyalgia Impact Questionnaire | 10 minutes
  Disease Severity and perceived physical function will be assessed with the "Revised Fibromyalgia Impact Questionnaire (FIQ-R)" consists of 21 questions in total. All questions in this questionnaire are rated on an 11-point numerical scale from 0 to 10, with 10 indicating the worst possible situation.
Short Form 12 (SF-12) | 10 minutes
  Quality of Life will be assessed with the SF-12 scale. SF-12, physical functionality (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functionality (1 item), emotional role (2 items) and mental health (2 items) and includes 8 sub-dimensions and 12 items in total. Both components range from 0 to 100, with a higher score representing better health.
Pain Catastrophe Scale (PCS) | 10 minutes
  Catastrophe will be assessed by the Pain Catastrophe Scale (PCS). The PCS is a 13-item self-report scale using a 5-point Likert scale (0-4).
The interview | 5 minutes
  Clinical history and patient interview will be done. The researcher will evaluate the symptoms of hypersensitivity based on the patient's clinical history. Besides, the researcher will evaluate whether the patient has increased sensitivity to odors, lights or sounds. Also, the researcher evaluates the patient's conditions such as fatigue, sleep disorders, and cognitive problems.

SECONDARY OUTCOMES:
Central Sensitization Inventory | 10 minute
  The Central Sensitization Inventory (CSI) aims to evaluate symptoms thought to be associated with nociplastic pain. It is also accepted as an effective scale used to evaluate patients with chronic pain who are also sensitive to the presence of neuropathic pain. The CSI consists 25 items exploring emotional and somatic disorders associated with CS. Each response is scored from 0 to 4, yielding a total score of 0 to 100 . A score of 40 or higher on the CSI means the presence of nociplastic pain.
Douleur Neuropathique 4 Questionnaire | 5 minutes
  The Douleur Neuropathique 4 (DN4) is one of the questionnaires that can be useful in diagnosing neuropathic pain. It has components of how the pain feels to the patient but also requires the examining health professional to assess whether there is reduced sensation (hypoaesthesia) to touch or pinprick and whether light brushing increases or causes pain (allodynia). The total score is calculated as the sum of the 10 items and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Saracoglu, P.hD., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Pamukkale University Hospitals, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided